CLINICAL TRIAL: NCT05094661
Title: Predictors of Non-invasive Respiratory Support Failure in COVID-19 Pneumonia
Acronym: RUTIROX
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Germans Trias i Pujol Hospital (Other)
Responsible Party: Principal Investigator, Irene Aldas, Principal Investigator, Respiratory Intermediate Care Unit., Germans Trias i Pujol Hospital
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: RUTIROX2021
Record Dates: First submitted 2021-04-22; First posted 2021-10-26 (Actual); Last update posted 2022-11-08 (Actual); Status verified 2022-08

CONDITIONS: Noninvasive Ventilation; Covid19; Distress; Respiratory Syndrome, Adult
Keywords: Covid19; Noninvasive ventilation; High flow oxygen
MeSH Terms: conditions — COVID-19; Acute Lung Injury

STUDY DESIGN:
Who Masked: Participant
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Non failure high flow oxygen therapy (No Intervention): The patient is treated with high flow oxygen system throughout the admission in the intermediate respiratory care unit
- Non-invasive ventilation (CPAP/BiPAP) (Active Comparator): If high flow support fails, the patients will be treated with non-invasive respiratory support.
  Interventions: Procedure: BiPAP; Procedure: CPAP

INTERVENTIONS:
Procedure: BiPAP — The patient recives respiratory support with bilevel positive airway pressure system until treatment improves or fails (needs intubation/dies).
  Arms: Non-invasive ventilation (CPAP/BiPAP)
Procedure: CPAP — The patient recives respiratory support with continuous positive airway pressure system until treatment improves or fails (needs intubation/dies).
  Arms: Non-invasive ventilation (CPAP/BiPAP)

SUMMARY:
The main objective of the current study is to search predictors of non-invasive respiratory support failure, like high -flow oxygen system (HFO) and pressure systems, Bilevel positive airway pressure (BiPAP) and continuous positive airway pressure (CPAP), in patients with acute hypoxemia produced by COVID-19 pneumonia.

In the first phase, we will do a retrospective review of the intermediate respiratory care unit activity from March to May 2020 in the target population. In the second phase development an interventional study. At admission all patients will be treated with HFS monitoring clinical variables like respiratory frequency, oxygen saturation, gasometer results and oxygen inspiration fraction. In case of HFO failure, the patients will be randomized to treatment with CPAP or BIPAP. The same clinical variables will be monitoring to analysis their prediction capacity of failure therapy, defined as mortality or need to intubation. The results will be adjusted comorbidity grade, age and initial severity pneumonia. Secondary objectives of study are 90 days mortality, functional recovery at 90 days and to realise a cost-effectiveness valuation of non-invasive respiratory supports in this disease.

DETAILED DESCRIPTION:
The purpose of the study

Pneumonia caused by the SARS Cov-2 coronavirus is a viral infectious disease that is characterized in some cases by the rapid and progressive respiratory failure of the respiratory system, being the most serious affectation and the one that marks the prognosis. Non-invasive breathing supports are therapies that help you breathe in severe respiratory failure. Therefore, monitoring of respiratory exhaustion should be carried out in all patients with SARS Cov-2 pneumonia. Within this follow-up, prognostic factors could be identified that help to assess with what probability the treatment with these supports may or may not be successful.

We will carry out a prospective, descriptive study at this center in order to assess respiratory clinical variables by telemetry recording and blood tests during follow-up.

To do this, we will carry out, during the follow-up of patients already diagnosed, or with a new diagnosis of SARS Cov-2 pneumonia and respiratory failure, who require non-invasive support therapy, an analysis on the first day of initiation of therapy, at 48 hours and at the end of this therapy, we will also continuously monitor vital signs while these therapies are used. We will compare the values obtained from patients who only require therapy with high-flow nasal cannulas and from patients who are not sufficient for this treatment and need non-invasive mechanical ventilation.

Participants in this study who do not have sufficient respiratory support with high-flow cannula therapy and feel exhausted, will be switched to non-invasive mechanical ventilation. Each patient will be randomly assigned to one of two possible settings: setting A (continuous pressure mechanical ventilation) or setting B (intermittent pressure mechanical ventilation). This decision is made because to date there are no scientifically proven differences in which configuration is best for the treatment of this disease. The data on the success of the therapies will be compared, understanding as failure the need for orotracheal intubation to perform invasive mechanical ventilation or death.

This research study has been approved by the Research Ethics Committee of the Germans Trias i Pujol University Hospital.

Study Procedures and Possible Risks and Discomforts Vital signs will be recorded during the time that non-invasive respiratory support therapy is performed continuously for the assessment of respiratory status. This does not pose any additional risk, since it is a non-invasive procedure and without exposure to ionizing radiation.

Between 3 and 5 tests will be carried out during the study, which are the same as those carried out in the usual clinical practice of this disease. They pose risks of pain due to puncture and extravasation of a blood vessel.

Participation in this study would not produce any discomfort except those derived from the non-invasive respiratory support therapies themselves. These are: epistaxis, runny nose, excessive noise in the treatment with high-flow cannulas and skin ulcers in the case of non-invasive mechanical ventilation. It does not imply an added risk to that of normal clinical practice for health since an additional intervention will not be carried out.

The information regarding your personal data (initials and medical record number) will be coded, a non-consecutive alphanumeric code will be assigned, which will be called the patient study code. This will only be known to the principal investigators, who will save this data using a password-protected Microsoft Excel file.

The clinical information collected for the study associated with your patient code will be stored in a Microsoft Excel type computer file located at the research center. The REDCAP form will be used for data collection. To access it, you will need a second password different from the first one. These data can only be re-identified by the study's principal investigators or by collaborators authorized by them. They will be used exclusively for the purposes specified here.

Voluntary participation and withdrawal You can freely decide whether or not you want to take part in this study, participation is completely voluntary. If you decide to participate, you still have the possibility to withdraw at any time, without having to give explanations, and without any penalty or negative consequences for you. If you change your mind regarding your samples or your data, you have the right to request their destruction or destruction. anonymization, through your doctor / researcher. However, you should know that the data obtained in the analyzes carried out up to that moment may be used for the purposes requested and may be kept in compliance with the corresponding legal obligations.

Participation in this study is not incompatible with participation in other clinical studies or trials.

Possible benefits No direct benefit is expected from your participation in the study. However, the information gained from this research project can contribute to medical advancement and could help other patients in the future. You will not receive any economic benefit for the transfer of the data provided, nor will you have rights over possible commercial benefits of the discoveries that may be achieved as a result of the research carried out.

Data protection and confidentiality

All information about your results will be treated strictly confidential. Your personal data will be identified by a code, so that it does not include information that can identify you, and only the research team will be able to relate that data to you. These data will be protected by password. These coded clinical data will be the ones that will be statistically analyzed to search for scientific findings that answer the questions proposed in this study. The analysis of this data will be carried out by the external company BUTLER SCIENTIFICS using Auto-discovery technology. This has signed a confidentiality and data treatment contract with the promoting center and the study researchers. This company will receive the data by means of a file with a password via email from the promoter center. BUTLER SCIENTIFCS in no case will know identifying data of the study participants. You may only make one research use for this study. You will not be able to trade or use the data for other purposes.

The Germans Trias i Pujol University Hospital - ICS Metropolitana Nord, as promoter and center where the study is carried out, assumes responsibility for data protection. Your personal data will be protected in accordance with the provisions of Organic Law 3/2018, of December 5, on the Protection of Personal Data and guarantee of digital rights and Regulation (EU) 2016/679 of the European Parliament and of the Council of 27 April 2016 on Data Protection (RGPD, having the right to access, rectify or cancel your data, and can limit the processing of data that are incorrect, request a copy or have the data that you have provided to a third party be transferred to To exercise your rights, contact the study's main researchers or collaborators whose data is specified at the end of this document. You can also contact the Data Protection Department of TIC Salut dpd@ticsalutsocial.cat . You also have the right to to contact the Data Protection Agency if you are not satisfied.

If the results of the study were subject to publication in scientific journals, personal data of the participants in this research will not be provided at any time.

Information on results In the event that you request it, at the end of the study and in accordance with article 27 of Law 14/2007 on Biomedical Research, information on the results of this research work may be provided to you

ELIGIBILITY:
Inclusion Criteria:

* Age ≥18 years.
* Severe hypoxemic respiratory failure (partial pressure of arterial oxygen/ fraction of inspired oxygen < 250 mmHg).
* Confirmed SARS-Cov2 infection.
* Radiological images compatible with pneumonia covid.

Exclusion Criteria:

* Hypoxemic respiratory failure secondary to a cause other than SARS-Cov2 pneumonia.
* Hypercapnic respiratory failure.
* Patient with criteria of orotracheal intubation at admission.
* Glasgow < 15
* Haemodynamic instability that needs drugs treatment
* Patients with swallowing problems that conditioned an aspiration pneumonia risk.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 135 (Actual)
Dates: Start 2021-02-18 (Actual); Primary Completion 2022-11-07 (Actual); Study Completion 2022-11-07 (Actual)

PRIMARY OUTCOMES:
Failure of High Flow Nasal Cannula | From the start of High Flow Nasal Cannula support to intubation and invasive ventilation or death at 30 days.
  The number of patients with respiratory work or desaturation at the beginning of therapy with high-flow nasal cannulas will be measured. This will be defined with desaturation below 90%, respiratory rate greater than 30 o pO2 below 60 despite receiving a maximum support of 60 liters per minute and with 100% FIO2.
Failure of Non Invasive Ventilation | From the start of CPAP or BIPAP to intubation and invasive ventilation or death at 30 days
  The number of patients with respiratory work or desaturation and who need orotracheal intubation or die will be measured. This will be defined with desaturation below 90%, respiratory rate above 30 o pO2 below 60 despite receiving a maximum pressure support and with 100% FIO2.

SECONDARY OUTCOMES:
90-day at home recovery | From the inclusion to 90 days after inclusion in the study.
  Compare the degree of pre-admission mMRC dyspnea with the degree of mMRC dyspnea 90 days after inclusion in the study.

CONTACTS AND LOCATIONS:
Overall Officials: Irene IA Aldás Criado, Principal Investigator — Germans Trias i Pujol Hospital
Locations (1):
- Germans TiPH, Barcelona, Spain

REFERENCES:
- [Background] Aliberti S, Radovanovic D, Billi F, Sotgiu G, Costanzo M, Pilocane T, Saderi L, Gramegna A, Rovellini A, Perotto L, Monzani V, Santus P, Blasi F. Helmet CPAP treatment in patients with COVID-19 pneumonia: a multicentre cohort study. Eur Respir J. 2020 Oct 15;56(4):2001935. doi: 10.1183/13993003.01935-2020. Print 2020 Oct. PMID 32747395
- [Background] Franco C, Facciolongo N, Tonelli R, Dongilli R, Vianello A, Pisani L, Scala R, Malerba M, Carlucci A, Negri EA, Spoladore G, Arcaro G, Tillio PA, Lastoria C, Schifino G, Tabbi L, Guidelli L, Guaraldi G, Ranieri VM, Clini E, Nava S. Feasibility and clinical impact of out-of-ICU noninvasive respiratory support in patients with COVID-19-related pneumonia. Eur Respir J. 2020 Nov 5;56(5):2002130. doi: 10.1183/13993003.02130-2020. Print 2020 Nov. PMID 32747398
- [Background] Frat JP, Thille AW, Mercat A, Girault C, Ragot S, Perbet S, Prat G, Boulain T, Morawiec E, Cottereau A, Devaquet J, Nseir S, Razazi K, Mira JP, Argaud L, Chakarian JC, Ricard JD, Wittebole X, Chevalier S, Herbland A, Fartoukh M, Constantin JM, Tonnelier JM, Pierrot M, Mathonnet A, Beduneau G, Deletage-Metreau C, Richard JC, Brochard L, Robert R; FLORALI Study Group; REVA Network. High-flow oxygen through nasal cannula in acute hypoxemic respiratory failure. N Engl J Med. 2015 Jun 4;372(23):2185-96. doi: 10.1056/NEJMoa1503326. Epub 2015 May 17. PMID 25981908
- [Background] Roca O, Caralt B, Messika J, Samper M, Sztrymf B, Hernandez G, Garcia-de-Acilu M, Frat JP, Masclans JR, Ricard JD. An Index Combining Respiratory Rate and Oxygenation to Predict Outcome of Nasal High-Flow Therapy. Am J Respir Crit Care Med. 2019 Jun 1;199(11):1368-1376. doi: 10.1164/rccm.201803-0589OC. PMID 30576221
- [Background] Carteaux G, Millan-Guilarte T, De Prost N, Razazi K, Abid S, Thille AW, Schortgen F, Brochard L, Brun-Buisson C, Mekontso Dessap A. Failure of Noninvasive Ventilation for De Novo Acute Hypoxemic Respiratory Failure: Role of Tidal Volume. Crit Care Med. 2016 Feb;44(2):282-90. doi: 10.1097/CCM.0000000000001379. PMID 26584191

DOCUMENTS (2):
  • Study Protocol and Statistical Analysis Plan (2021-01-21): https://cdn.clinicaltrials.gov/large-docs/61/NCT05094661/Prot_SAP_002.pdf
  • Informed Consent Form (2021-01-21): https://cdn.clinicaltrials.gov/large-docs/61/NCT05094661/ICF_001.pdf